CLINICAL TRIAL: NCT04806438
Title: Airway Nerve Block Versus Nebulization by Lignocaine During Diagnostic Flexible Bronchoscopy Under Moderate Sedation. A Randomized Controlled Trial
Brief Title: Airway Nerve Block Versus Nebulization by Lignocaine During Diagnostic Flexible Bronchoscopy Under Moderate Sedation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R128/2020
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (nebulized lignocaine group) (Active Comparator): Patients will receive 5 ml of 10% lignocaine by air driven jet nebulizer for 20 min
  Interventions: Other: Group A
- Group B (nerve block group) (Active Comparator): Patients will receive bilateral superior laryngeal nerve block and transtracheal instillation of 4 ml of 2% lignocaine, along with viscous xylocaine gargles twice.
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Patient will receive 5 ml of 10% lignocaine by air driven jet nebulizer for 20 min
  Other Names: Lignocaine nebulizer
  Arms: Group A (nebulized lignocaine group)
Other: Group B — Patients will receive bilateral superior laryngeal nerve block and transtracheal instillation of 4 ml of 2% lignocaine, along with viscous xylocaine gargles twice
  Other Names: Airway nerve block
  Arms: Group B (nerve block group)

SUMMARY:
To compare the effectiveness of nebulization versus airway nerve block technique to achieve upper airway anesthesia for diagnostic fiberoptic bronchoscopy under moderate sedation.

DETAILED DESCRIPTION:
Randomization was done using computer generated tables of random numbers:

Group A (nebulized lignocaine group) as a control group (n = 60) received 5 ml of 10% lignocaine by air driven jet nebulizer for 20 min .

Group B (nerve block group) (n = 60) received bilateral superior laryngeal nerve block and trans-tracheal instillation of 4 ml of 2% lignocaine, along with viscous xylocaine gargles twice.

Patient tolerance was assessed using the Global Tolerance Score, based on a visual analogue scale ( VAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for diagnostic fiberoptic procedures such as broncho-alveolar lavage, endobronchial or transbronchial biopsies, or brush cytology.

Exclusion Criteria:

* Patients less than 21yrs old and patients more than 70 yrs old.
* Severe respiratory failure (pH < 7.35, partial arterial oxygen pressure <55 mmHg despite supplemental oxygen).
* Upper airway surgery or radiation, allergy to lidocaine, Propofol or midazolam, or bleeding disorder.
* Hemodynamic instable patient or patient decompensated heart failure.
* Epileptic patients, severe neurological or psychiatric disorder.
* Patients requiring cryo-biopsy or endobronchial ultrasound because these procedures are performed under deep sedation including fiberoptic intubation.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-21 (Estimated); Primary Completion 2021-06-21 (Estimated); Study Completion 2021-07-21 (Estimated)

PRIMARY OUTCOMES:
Global Tolerance Score | First two hours in the postoperative period
  The Tolerance Score, defined as the arithmetic mean of global tolerance visual analogue score (VAS)and the mean of scores for the 4 specific sensations, was calculated.